CLINICAL TRIAL: NCT04823286
Title: REVID +: Integrated Patient Care Intradialysis Programme in Hemodialysis Through a Virtual Health Platform (GoodRENal.eu)
Brief Title: Integrated Patient Care Intradialysis Programme in Hemodialysis Through a Virtual Health Platform
Acronym: GoodRENal
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de Manises (Other); Universitat Politècnica de València (Other); University of Valencia (Other); Karolinska Institutet (Other); Skane University Hospital (Other); KU Leuven (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-064-1
Record Dates: First submitted 2021-01-28; First posted 2021-03-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease; Hemodialysis-Induced Symptom; Chronic Kidney Diseases
Keywords: exercise; physical function; health related quality of life; nutrition; psychological wellbeing
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups, intradialysis virtual reality platform or usual care
Who Masked: Investigator, Outcomes Assessor
Masking Description: A team of assessors, different to the researchers implementing the exercise, will record all dependent variables. A blind researcher will randomize participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality health platform during hemodialysis (Experimental): During 12 weeks subjects will use a VR platform during hemodialysis. The intervention will be virtual reality exercise, nutritional advice and psychological wellbeing support plus cognitive training.
  Interventions: Other: Virtual reality health platform during hemodialysis
- Control group-usual care (No Intervention): During 12 weeks subjects will carry on with the usual care in the hemodialysis unit

INTERVENTIONS:
Other: Virtual reality health platform during hemodialysis — Subjects will play a virtual reality game specially adapted for subjects undertaking hemodialysis. The game will also aim at providing nutritional advice, and improving psychological wellbeing and cognitive function.
  Arms: Virtual reality health platform during hemodialysis

SUMMARY:
There is wide evidence regarding the weak points of end-stage Chronic kidney disease (CKD) patients in hemodialysis, and they include three intervention aspects: exercise, nutrition and psychological support. Evidence shows that exercise for patients in hemodialysis results in increased survival rate, functional capacity, strength and health-related quality of life.

Additionally, different studies have shown the benefits of psychological interventions and the positive effect of educational programs on nutritional care for patients in hemodialysis.

Despite the well-known benefits of exercise, this kind of programs are not being implemented in the routine clinical care of hemodialysis patients.

Thus, the GoodRENal project aims to promote healthy lifestyles among dialysis patients in a holistic approach that combines exercise, nutrition and psychological wellbeing plus cognitive functioning addressing adult learners. The project will, in phase 1, explore barriers and facilitators of patients, carers and health professionals towards healthy lifestyle (physical activity, nutrition and psychological well being). In phase 2, the project will develop a health virtual platform including these three dimensions of cares. In summary, the project outputs will be:

1. A didactic content in a modular platform to create an educational program for integrated treatments in patients with dialysis
2. A guideline to promote healthy lifestyles among dialysis patients for health care providers
3. A guideline to promote e healthy lifestyles among dialysis patients for patients and formal - nonformal carers

DETAILED DESCRIPTION:
CKD stage 5D, has a high incidence, 100-200 people per million, and high prevalence, 750-1500 per million. More than 40-50% are above 65 years old, with a lower rate in women but with higher frailty than men. This cohort presents high comorbidity, malnutrition, sedentary behavior, low health-related quality of life, frailty and high dependency levels. Mortality risk is close to 15% per year. Cardiovascular disease is the main cause of death in end-stage CKD. It is also a high risk factor for peripheral artery disease and lower limbs amputation.

Supporting this cohort results in high direct and indirect costs. Additionally, these patients present high anxiety and depression rates. Comorbidity between depression and somatic illness leads to a significant increase of the illness load since there is higher symptomatology, higher morbidity, higher health costs, and worse functioning and quality of life. Current evidence suggests a bidirectional relationship between depression and medical illness. Mechanisms suggested explaining this complex relationship would include both biological and behavioral aspects. Depression is also associated with the worst adherence to treatment of comorbid patients.

There is wide evidence regarding the weak points of end-stage CKD patients in hemodialysis, and they include three intervention aspects: exercise, nutrition and psychological support. Evidence shows that exercise for patients in hemodialysis results in increased survival rate, functional capacity, strength, and health-related quality of life. Additionally, different studies have shown the benefits of psychological interventions and the positive effect of educational programs on nutritional care for patients in hemodialysis. Several combined interventions have been implemented leading to heterogeneous results.

Despite the well-known benefits of exercise, this kind of programs are not being implemented in the routine clinical care of hemodialysis patients. Patients' lack of interest regarding participation in exercise programs, time constraints, and lack of knowledge by health professionals at the hemodialysis units, are some of the factors underpinning the low implementation rate of intradialysis exercise programs.

Virtual reality (VR) refers to computer-generated interactive simulation that offers users the opportunity to participate in environments that look like objects and events of the real world.

VR exercise has been successfully implemented in neuro-rehabilitation, resulting in better balance, gait, and mobility in cerebrovascular accidents, multiple sclerosis, Guillain-Barre syndrome, and Parkinson's disease. Few studies have explored the impact of VR exercise in renal rehabilitation. Three of the partners (Universidad Cardenal Herrera-CEU, Universitat Politècnica de Valéncia, and Hospital de Manises) have implemented two randomized trials of non-immersive VR exercise intradialysis. Currently, those partners are developing a third trial with this technology and they have verified that this type of exercise has good tolerance and high adherence rates. Additionally, it has a positive impact on strength, functional capacity, physical activity level, and health-related quality of life.

Until now, the most traditional way to assess and implement psychological and psycho-educative treatments has been 'face to face'. Nevertheless, more than 50% of people suffering from depression are not being treated appropriately. This is why alternative treatment models to assess and treat are being implemented, and technology (as the internet) is an option to increase the number of patients that can be treated. Additionally, few studies have explored technology as a means to educate renal patients regarding nutrition or psychological health.

Thus, the hypothesis of the present study is that a health virtual platform designed for holistic treatment of patients undertaking hemodialysis will result in health benefits for this cohort, regarding physical activity, nutritional and psychological health. The platform will be designed according to the aims highlighted by experts, barriers, and needs of end-stage CKD patients and their caregivers. As mentioned above, end-stage chronic kidney disease patients have high comorbidity, malnutrition, sedentarism, low health-related quality of life, low physical function, frailty, and high dependency levels. So they rely on non-formal caregivers for their activities of daily living. This cohort presents high anxiety and depression levels and the combination of somatic disease plus depression results in higher symptoms, higher comorbidity, higher health resources, and worst quality of life. Besides, there is a bidirectional relationship between depression and disease, and depression is associated with lower adherence to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients on hemodialysis medically stable
* Ability to walk to walk at least a few steps, even if walking aids like canes or a walker ar needed
* Life expectancy greater than 6 months

Exclusion Criteria:

* Myocardial infarction in the previous 6 weeks
* Angina unstable on exercise or at rest
* Brain injury derived from a cardiovascular problem. Cerebral vascular disease such as stroke in the last 6 months or with relevant sequelae in lower limb mobility presenting hemiparesia.
* Life expectancy less than 6 months
* Cognitive impairment
* Language barriers
* Illiteracy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline distance walked assessed by the 6 minutes walk test at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  More meters walked in 6 minutes mean a better walking capacity

SECONDARY OUTCOMES:
Change from baseline health-related quality of life assessed by the Short Form 36 questionnaire at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The short form 36 gives data on 8 subscales and 2 components, higher score mean better health-related quality of life The scores range from 0 to 100, with 100 indicating optimal health and 0 reflecting very poor health.
Change from baseline stance from a chair capacity assessed by the sit to stand 10 at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Time in seconds to perform 10 sit to stand repetitions. A decrease in the time to perform the test means better functional capacity to stand up from a chair
Change from baseline usual gait speed assessed by a 4 meters gait speed test at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Speed in m/s to cover 4 meters at normal speed. An increase in speed to perform the test means better gait speed
Change from baseline handgrip strength assessed by a handgrip dinamometer at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Bilateral handgrip strength measured in kilograms. An increase in handgrip strength means better strength
Change from baseline lower limbs strength assessed by a dinamometer at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Bilateral lower limbs muscle strength measured in kilograms. An increase in strength means better strength
Change from baseline physical activity level assessed by the human activity profile questionnaire, average activity score at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The average activity score of the human activity profile questionnaire ranges from 0 to 94. . A higher score means a higher physical activity level
Change from baseline physical activity level assessed by the international physical activity questionnaire at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The score of the international physical activity questionnaire will be recorded in MET-minutes/week. A higher score means a higher physical activity level
Percentage of sessions performed from te sessions offered to measure adherence to the educational program | After 12 weeks of intervention
  Calculation will be the result of sessions performed/sessions offered
Healthcare resources expenditure and costs | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Total amount in euros spent on external consultations, laboratory tests, radiology tests, hospital pharmacy, emergency department healthcare provision, and hospitalisation.
Change from baseline lean body mass assessed by the bioimpedance spectroscopy at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Lean body mass is a surrogate of muscle mass in kilograms. Increase in lean body mass means increase in muscle mass
Change from baseline qualitative assessment in food intake assessed by the Short form food questionnaire at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Qualitative assessment of food intake Short form food questionnaire. Improvement in the dietary quality
Change from baseline nutritional status assessed by the 7 point Subjective Global Assessment at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  7 point subjective global assessment scores from 1 to 7, the higher the score the better nutritional status
Change from baseline cognitive function assessed by the Mini-mental State at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The maximum MMSE score is 30 points. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.
Change from baseline Anxiety assessed by the Hospital Anxiety and Depression Scale at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Scores obtained between 0 and 21. The higher the score obtained, the higher the level of anxiety and depression.
Change from baseline positive and negative emotions assessed by Positive and Negative Affect Schedule Scale (PANAS) at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  It includes 2 subscales (positive affect and negative affect) with 10 items each. Each subscale can contain scores between 10 and 50. The higher the score obtained, the greater the presence of a particular affect.
Change from baseline depression assessed by the Beck Depression Inventory (BDI) at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The scores range from 0 to 63 points. The higher the score, the greater the severity of depressive symptoms. Four groups are established according to the total score: 0-13, minimal depression; 14-19, mild depression; 20-28, moderate depression; and 29-63, severe depression.
Change from baseline anxiety assessed by the State Trait Anxiety Inventory (STAI) at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Scale composed of 2 subscales. The range of scores for both subscales is between 0 and 60 points so that higher scores reflect greater anxiety.
Change from baseline perceived stress assessed by the Perceived Stress Scale (PSS) at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Scores obtained in a range of 0 to 56 points. The higher the score obtained, the higher the level of perceived stress.
Change from baseline cognitive state assessed by the Montreal Cognitive Assessment (MoCA)at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Scores on the MoCA assessment range from 0 to 30. A score of 26 and above is considered normal.
Change from baseline attention level assessed by the Trail Making Test (TMT) at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  Scoring is based on time taken to complete the test, with lower scores being better.
Change from baseline memory assessed by the Wechsler-IV Memory Scale at 12 weeks | Baseline, after 12 weeks of intervention, 12 weeks follow-up after the end of the intervention
  The correction system allows obtaining scalar scores, indices, centiles and confidence intervals, in order to achieve a more flexible interpretation. It is interpreted on the basis of scales. The Spanish scales have been elaborated from a sample of almost 900 subjects aged between16 and 90 years.

CONTACTS AND LOCATIONS:
Overall Officials: Eva SEGURA-ORTÍ, Principal Investigator — Universidad CEU Cardenal Herrera, UCH CEU
Locations (8):
- KU Leuven, Leuven, Belgium
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Spain (4):
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital de Manises, Manises, Valencia
  - Universitat de Valencia, Valencia, Valencia
  - Universitat Politécnica de Valéncia, Valencia, Valencia
- Sweden (2):
  - Skane Univeristy Hospital, Lund
  - Karolinska Institute, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segura-Orti E, Gordon PL, Doyle JW, Johansen KL. Correlates of Physical Functioning and Performance Across the Spectrum of Kidney Function. Clin Nurs Res. 2018 Jun;27(5):579-596. doi: 10.1177/1054773816689282. Epub 2017 Jan 23. PMID 28114792
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Background] Segura-Orti E, Johansen KL. Exercise in end-stage renal disease. Semin Dial. 2010 Jul-Aug;23(4):422-30. doi: 10.1111/j.1525-139X.2010.00766.x. PMID 20701722
- [Background] Segura-Orti E. [Exercise in haemodyalisis patients: a literature systematic review]. Nefrologia. 2010;30(2):236-46. doi: 10.3265/Nefrologia.pre2010.Jan.10229. Epub 2010 Jan 21. Spanish. PMID 20098466
- [Background] Segura-Orti E, Kouidi E, Lison JF. Effect of resistance exercise during hemodialysis on physical function and quality of life: randomized controlled trial. Clin Nephrol. 2009 May;71(5):527-37. doi: 10.5414/cnp71527. PMID 19473613
- [Background] Segura-Orti E, Rodilla-Alama V, Lison JF. [Physiotherapy during hemodialysis: results of a progressive resistance-training programme]. Nefrologia. 2008;28(1):67-72. Spanish. PMID 18336134